CLINICAL TRIAL: NCT04849572
Title: Sleep Well Live Well (SWELL) Pilot Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2103262999
Record Dates: First submitted 2021-04-13; First posted 2021-04-19 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2023-08

CONDITIONS: Sleep Hygiene
MeSH Terms: conditions — Sleep Hygiene

STUDY DESIGN:
Intervention Model Description: This is a permuted block randomization study to assess the efficacy of the new intervention and the primary outcome variable is the sleep time. A total of 100 subjects (50 per group) will be randomized to each treatment group, stratified by gender. The first group will receive the intervention and be enrolled into the trial after the run-in period and the baseline data collection, and the second group will receive the intervention at 6 weeks after trial start.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep Education (Active Comparator): Also referred to as Arm 1. Arm 1 receives sleep education initially.
  Interventions: Behavioral: Sleep Education
- Delayed Sleep Education (Active Comparator): Also referred to Arm 2. Arm 2 receives no initial sleep education.
  Interventions: Behavioral: Delayed Sleep Education

INTERVENTIONS:
Behavioral: Sleep Education — * Week 1-2: All 100 participants will have sleep parameters recorded as baseline for the first two weeks.
  * Week 3: 50 participants (Arm 1) will watch a 10 to 20 minute sleep hygiene video followed by a post-test questionnaire to confirm participation and understanding.
  * Week 5: Arm 1 will again view the educational video at week 5
  * Week 6-8: Baseline sleep data on all participants will be downloaded for review and the PSQI questionnaire administered for both groups. Participants will be also be asked if they underwent any major health crisis during the study period which may have impacted their sleep (hospitalization, significant medication changes which they believe impacted sleep, any use of illicit drugs during the study periods or significant increase in alcohol consumption (e.g., doubling).
  * Week 9: Arm 1 will continue re-education
  * Week 11: Arm 1 continues education
  * Week 12-14: Data from Oura ring will be downloaded and PSQI administered to both groups.
  Arms: Sleep Education
Behavioral: Delayed Sleep Education — * Week 1-2: All 100 participants will have sleep parameters recorded as baseline for the first two weeks.
  * Week 3: 50 participants (Arm 2) will be controls with no education.
  * Week 6-8: Baseline sleep data on all participants will be downloaded for review and the PSQI questionnaire administered for both groups. Participants will be also be asked if they underwent any major health crisis during the study period which may have impacted their sleep (hospitalization, significant medication changes which they believe impacted sleep, any use of illicit drugs during the study periods or significant increase in alcohol consumption (e.g., doubling).
  * Week 9: Arm 2 will join in for video education along with post-test
  * Week 11: Arm 2 will undergo reeducation with post-test for 20 mins
  * Week 12-14: Data from Oura ring will be downloaded and PSQI administered to both groups.
  Arms: Delayed Sleep Education

SUMMARY:
This will be a 12 week randomized control trial of sleep hygiene education vs. no education with a cross-over to the active intervention after 6 weeks. Primary and secondary outcomes will be assessed before and after a 10-20 minute sleep hygiene video (intervention).

DETAILED DESCRIPTION:
The primary aim of this study is to assess if sleep hygiene education increases sleep duration and sleep quality in an Appalachian community. To accomplish these aims, the investigators will assess changes in sleep duration by the Oura ring and the PSQI and Epworth Sleepiness Scale (ESS). Secondary aims are to determine whether sleep hygiene education decreases heart rate variability measured by the Oura ring and improves alertness as assessed by psychomotor vigilance testing (PVT). Potential participants will be recruited via brochures, poster displays and on-line media to participate in the study. Those eligible will be asked to complete a questionnaire to record baseline demographics. The data collected will be demographic information, presence of chronic medical conditions, validated sleep questionnaires, PVT results and Oura ring (https://ouraring.com/) output. A total of 100 subjects (50 per group) will be randomized to each treatment group, stratified by gender. The first group will receive the intervention and be enrolled into the trial after the run-in period and the baseline data collection, and the second group will receive the intervention at 6 weeks after trial start. Each subject (in both groups) will have pre- and post-intervention data in this study. Therefore, the "real" control in this study is the subject himself/herself (after taking the difference), which will minimize any confounding factors/effect; If the investigators assume that more education duration will result in more benefit, the investigators have a chance to assess a dose-response curve ("dosage" = education duration). The investigators will fit a mixed-effects model with duration as a fixed effect, adjusting for potential confounding variables if any.

ELIGIBILITY:
Inclusion Criteria:

* Reside in Harrison County of West Virginia
* Ability to read and understand English
* Ability to provide informed consent

Exclusion Criteria:

* Inability to read and understand English
* Inability or unwillingness to provide informed consent
* Presence of sleep apnea
* Depression
* Severe insomnia
* Using prescription sleeping medication or narcotics
* Acute illness including stroke, heart attack, heart failure or pneumonia with or without COVID-19 infection requiring hospital admission within the last 8 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Efforts will be made to have 50% female participation to reflect the gender ratio in Appalachia. A total of 100 subjects (50 per group) will be randomized to each treatment group, stratified by gender.
Enrollment: 106 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2022-05-06 (Actual); Study Completion 2022-05-06 (Actual)

PRIMARY OUTCOMES:
Difference in total sleep time | 6 Weeks
  A 20 minute or more difference in total sleep time between Arm 1 (sleep education) and Arm 2 (no initial sleep education).
Change in the ESS in Arm 1 (≥2 points) | 6 Weeks
  The Epworth Sleepiness Scale (ESS) is widely used in the field of sleep medicine as a subjective measure of a patient's sleepiness. The test is a list of eight situations in which the subjects rate their tendency to become sleepy on a scale of 0, no chance of dozing, to 3, high chance of dozing. When the subjects finish the test, add up the values of the responses. The subjects total score is based on a scale of 0 to 24. The scale estimates whether the subjects are experiencing excessive sleepiness that possibly requires medical attention.
Change in PSQI at 6 weeks in Arm 1 (≥3 points) | 6 Weeks
  The Pittsburgh Sleep Quality Index (PSQI) contains 19 self-rated questions and 5 questions rated by the bed partner or roommate (if one is available). Only self-rated questions are included in the scoring. The 19 self-rated items are combined to form seven "component" scores, each of which has a range of 0-3 points. In all cases, a score of "O" indicates no difficulty, while a score of "3" indicates severe difficulty. The seven component scores are then added to yield one "global" score, with a range of 0-21 points, "O" indicating no difficulty and "21 " indicating severe difficulties in all areas.

SECONDARY OUTCOMES:
Change in total sleep time | 6 weeks after sleep education
  Change in total sleep time variability (> 1 hour) in both groups. Changes in sleep duration will be assessed by the Oura ring, a novel sleep monitoring device.
Change in daytime alertness as measured by psychomotor vigilance testing (PVT) in both groups | 6 weeks after sleep education
  The primary outcome measures of PVT performance, lapses, are defined as reaction times exceeding 500 msec or failure to react. The PVT lapses are believed to represent perceptual, processing, or executive failures in the central nervous system (CNS).
Change in heart rate variability in both groups | 6 weeks after sleep education
  Measured by the Oura Ring

CONTACTS AND LOCATIONS:
Locations (1):
- West Virginia University, Morgantown, West Virginia, United States

REFERENCES:
- [Derived] Sharma S, Stansbury R, Ramadan J, Rojas E, Finomore V, Pham C, Quan SF, Wen S. Sleep well and live well: Impact of sleep hygiene intervention on sleep duration in a rural community: A randomized controlled trial (THE SWELL STUDY). J Rural Health. 2025 Jan;41(1):e70002. doi: 10.1111/jrh.70002. PMID 39930329